CLINICAL TRIAL: NCT04995211
Title: Validity and Reliability of Commercially Available Metabolic Carts
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Associate Executive Director for Clinical Science, Pennington Biomedical Research Center
Other Study IDs: PBRC2020-036
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Metabolism and Nutrition Disorder
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Assessment of resting energy expenditure — We will assess the resting metabolic rate and respiratory exchange ratio of twenty healthy adults, with every metabolic cart on two days in the morning. The assessment will last 30 minutes on each metabolic cart, with 15-minute breaks between measurements. The order of the metabolic carts will be randomly selected and replicated the second day.

SUMMARY:
The validity (by alcohol burning and gas infusions) and reliability (day-to-day variability in healthy subjects) of six metabolic carts will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female.
* Age 18-65 y.
* BMI between 18.5 kg/m2 and 40 kg/m2 (inclusive).
* Are willing to fast and not consume non-caloric stimulant for 10h before the assessments, and during the stay in the center.
* Are willing to avoid moderate or vigorous physical activity during 24h before the visits.

Exclusion Criteria:

* Smoking or use of tobacco products within the last 3 months
* Diagnosed with diabetes.
* Previous bariatric surgery (or other surgeries) for obesity or weight loss.
* Use of medications affecting metabolism or sleep.
* History of neurological disease.
* History of cardiovascular disease, including hypertension, or other chronic diseases.
* Pregnant, planning to become pregnant, or breastfeeding
* Claustrophobia impeding to stay calm under a plastic canopy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Resting metabolic rate | 30 minutes
  Indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States